CLINICAL TRIAL: NCT06882499
Title: Stereotactic Ablative Body Radiotherapy (SABR) with Maintenance of Systemic Therapy Versus Physicians' Choice of Systemic Therapy for Oligoprogressive ER-positive, Her-2 Negative Breast Cancer II
Acronym: AVATAR II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Monash Health (Other); Monash Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMC105165 (24/143)
Record Dates: First submitted 2024-12-08; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer, Metastatic; Metastatic Breast Cancer
Keywords: ER-positive, HER2-negative; selective estrogen receptor degrader; endocrine therapy; aromatase inhibitor; CDK 4/6 inhibitor; SABR; oligoprogression; oligometastases; oligometastatic; sbrt
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SABR to all known sites of oligoprogressive disease with continuation of first line therapy (Experimental): SABR to all known sites of oligoprogressive disease with continuation of first line therapy ET + CDK4/6i
  Interventions: Radiation: Stereotactic Ablative Radiotherapy
- Physician's choice of systemic treatment (Active Comparator): Physician's choice of systemic treatment does not mandate a change in systemic therapy, however, SABR is not permitted for management in this arm
  Interventions: Other: Physician's choice of systemic treatment

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy — Stereotactic Ablative Radiotherapy
  Arms: SABR to all known sites of oligoprogressive disease with continuation of first line therapy
Other: Physician's choice of systemic treatment — Physician's choice of systemic therapy does not mandate a change in systemic therapy, however, SABR is not permitted for management in this arm
  Arms: Physician's choice of systemic treatment

SUMMARY:
The goal of this clinical trial is to assess Stereotactic Ablative Radiotherapy (SABR) as a method to delay a change in systemic therapy in patients with oligoprogressive ER-positive, HER2-negative advanced breast cancer. The main question it aims to answer is to assess whether the addition of SABR to continuation of first line endocrine therapy and CDK 4/6 inhibitor (Arm A) to patients with oligoprogressive ER-positive, HER2-negative advanced breast cancer could have longer time to strategy failure (TSF) in comparison to physician choice of systemic treatment (Arm B) in patients who had progressed first line.

The treatment strategy in Arm A is to maintain patients on current endocrine therapy and CDK 4/6 inhibitor, controlling localised progressing sites of disease with SABR. Treatment strategy in Arm B is to maintain disease control with physician's choice of systemic therapy alone.

DETAILED DESCRIPTION:
AVATAR II is a phase II multicentre open label, randomised trial. Following informed consent, eligible patients with ER-positive, HER2-negative advanced breast cancer receiving an ET (either AI or selective estrogen receptor degrader in combination with a CDK 4/6 inhibitor with newly diagnosed OPD amenable to SABR will be randomised to either:

Arm A: SABR to all known sites of OPD with continuation of first line therapy ET and CDK 4/6 inhibitor Arm B: Physician's choice of systemic treatment

Patients must have evidence of radiological response to ET and CDK 4/6 inhibitor for a minimum of six months prior to randomisation (defined as either stable disease or partial response).

All patients will be followed up for 3 years after the last patient has been randomised.

ELIGIBILITY:
INCLUSION CRITERIA

Patients will be eligible for inclusion in this trial if all the following criteria apply:

1. Patient has signed the AVATAR-II Patient Information and Consent Form (PICF)
2. Male or female, ≥ 18 years of age at the time signing consent
3. Patients with histologically proven ER-positive, HER2-negative advanced breast cancer receiving an ET in combination with a CDK 4/6 inhibitor. Biopsy of metastatic disease if technically feasible but not mandatory
4. Patients must have evidence of extracranial metastatic disease, with no evidence of uncontrolled intracranial metastases
5. Patients must have evidence of radiological response to ET and CDK 4/6 inhibitor for a minimum of six months prior to randomisation (defined as either stable disease or partial response) Note: Patient must have ongoing stability/response in at least one lesion at the time of randomisation.
6. Evidence of new or existing OPD, as determined by the Investigator and defined according to RECIST1.1 (33), via CT on a per-lesion basis (between 1-5 metastases, including the primary) as follows:

   * At least a 20% increase in the diameter of a lesion, taking as reference the smallest diameter on a previous CT scan with an absolute increase of at least 5 mm
   * Appearance of a new lesion(s) Note: A new lesion can be identified using various imaging modalities, such as PET-CT or WBBS, as long as the lesion is visible on serial CT scans.
7. For patients with liver or lung metastases, maximum of 3 oligoprogressive lesions in single organ
8. All OPD must be amenable to SABR, as per the radiotherapy guidelines in section 11.1 and Appendix 4 and 5
9. ECOG performance status 0-2
10. Life expectancy ≥ 6 months
11. Clinician and patient are willing to continue current line of therapy
12. Patient is able to complete QoL questionnaires, and other assessments required as part of the study

EXCLUSION CRITERIA

Patients will not be eligible for inclusion in this trial if any of the following criteria apply:

1. Is pregnant or lactating at the time of randomisation
2. Evidence of more than one clone of metastatic disease e.g., a patient with both ER-positive and triple negative clones of disease And ER-negative and/or HER2-positive disease would be excluded from the study
3. Evidence of leptomeningeal disease
4. Evidence of malignant cord compression
5. Evidence of lesion within femoral bone requiring surgical fixation
6. Patients with risk of bone fracture are not candidate for SABR (Appendix 4 and 5)
7. Previous chemotherapy for metastatic disease Note: chemotherapy for primary breast cancer is allowed
8. Contraindications to radiotherapy
9. Any condition deeming the patient unsuitable to comply with the study
10. Substantial overlap with previously treated area. Reirradiation is permitted with the condition that the combined plan adheres to the specific dose constraints outlined in this protocol. It is advised to use biological effective dose (BED) calculations to correlate previous doses with the tolerance doses documented below

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2032-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause assessed until withdrawal of consent, death, or 3 years after the last patient has been randomised, whichever is earlier.
  The primary endpoint of this study is to measure the Time to Strategy Failure between Arm A and Arm B.
  Treatment strategy failure is defined as time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause.
  Progression, as determined by the Investigator, will be defined according to the Response Evaluation Criteria in Solid Tumors, Version 1.1. (RECIST1.1; Appendix 2) (33) The treatment strategy in Arm A is to maintain patients on current ET and CDK 4/6 inhibitor, controlling localised progressing sites of disease with SABR. Treatment strategy in Arm B is to maintain disease control with physician's choice systemic therapy alone.

SECONDARY OUTCOMES:
Secondary Objective 1 | Time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause assessed until withdrawal of consent, death, or 3 years after the last patient has been randomised, whichever is earlier.
  To compare PFS; PFS is assessed from randomisation to the date of the first evidence of progression or death by any cause. A patient will be considered to have progressed if there is evidence on progression according to RECIST1.1 or clinical progression
Secondary Objective 2 | Time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause assessed until withdrawal of consent, death, or 3 years after the last patient has been randomised, whichever is earlier.
  To compare progression-free survival 2 (PFS-2); PFS-2 is assessed from randomisation to the date of progression on next line of systemic anti-cancer treatment or death by any cause.
Secondary Objective 3 | Time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause assessed until withdrawal of consent, death, or 3 years after the last patient has been randomised, whichever is earlier.
  To compare PFS of next line of treatment (2nd PFS); 2nd PFS is assessed from failure of treatment strategy to progression on next line of systemic anti-cancer treatment or date of death by any cause.
Secondary Objective 4 | Time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause assessed until withdrawal of consent, death, or 3 years after the last patient has been randomised, whichever is earlier.
  To compare OS; OS is assessed from randomisation to the date of death by any cause.
Secondary Objective 5 | Time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause assessed until withdrawal of consent, death, or 3 years after the last patient has been randomised, whichever is earlier.
  To compare treatment related adverse events (TRAEs); TRAEs are adverse events assessed using the Common Terminology for Adverse Events Version 5.0 (CTCAE v5.0) considered possibly, probably, or definitely related to treatment (systemic therapy or SABR)
Secondary Objective 6 | Time from randomisation to progression of disease resulting in a failure of treatment strategy or death by any cause assessed until withdrawal of consent, death, or 3 years after the last patient has been randomised, whichever is earlier.
  To compare the QoL using the FACT-B total score: Area under the curve (AUC) of the FACT-B Total score from baseline to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Steven David, Principal Investigator — Peter MacCallum Cancer Centre, Australia

IPD SHARING:
Plan to Share IPD: No
Not contractually obliged but it may be considered

REFERENCES:
- [Background] Alomran R, White M, Bruce M, Bressel M, Roache S, Karroum L, Hanna GG, Siva S, Goel S, David S. Stereotactic radiotherapy for oligoprogressive ER-positive breast cancer (AVATAR). BMC Cancer. 2021 Mar 23;21(1):303. doi: 10.1186/s12885-021-08042-w. PMID 33757458
- [Background] David SP, Siva S, Bressel M, Tan J, Hanna GG, Alomran RK, et al. Stereotactic Ablative Body Radiotherapy (SABR) for Oligoprogressive ER-Positive Breast Cancer (AVATAR): A Phase II Prospective Multicenter Trial. International journal of radiation oncology, biology, physics. 2023;117(4):e6-e.
- [Background] Kelly P, Ma Z, Baidas S, Moroose R, Shah N, Dagan R, Mamounas E, Rineer J. Patterns of Progression in Metastatic Estrogen Receptor Positive Breast Cancer: An Argument for Local Therapy. Int J Breast Cancer. 2017;2017:1367159. doi: 10.1155/2017/1367159. Epub 2017 Sep 25. PMID 29147583
- [Background] Patel PH, Palma D, McDonald F, Tree AC. The Dandelion Dilemma Revisited for Oligoprogression: Treat the Whole Lawn or Weed Selectively? Clin Oncol (R Coll Radiol). 2019 Dec;31(12):824-833. doi: 10.1016/j.clon.2019.05.015. Epub 2019 Jun 8. PMID 31182289
- [Background] Cheung P. Stereotactic body radiotherapy for oligoprogressive cancer. Br J Radiol. 2016 Oct;89(1066):20160251. doi: 10.1259/bjr.20160251. Epub 2016 Aug 24. PMID 27556349
- [Background] Chan OSH, Lee VHF, Mok TSK, Mo F, Chang ATY, Yeung RMW. The Role of Radiotherapy in Epidermal Growth Factor Receptor Mutation-positive Patients with Oligoprogression: A Matched-cohort Analysis. Clin Oncol (R Coll Radiol). 2017 Sep;29(9):568-575. doi: 10.1016/j.clon.2017.04.035. Epub 2017 May 9. PMID 28499791
- [Background] Weickhardt AJ, Scheier B, Burke JM, Gan G, Lu X, Bunn PA Jr, Aisner DL, Gaspar LE, Kavanagh BD, Doebele RC, Camidge DR. Local ablative therapy of oligoprogressive disease prolongs disease control by tyrosine kinase inhibitors in oncogene-addicted non-small-cell lung cancer. J Thorac Oncol. 2012 Dec;7(12):1807-1814. doi: 10.1097/JTO.0b013e3182745948. PMID 23154552
- [Background] Xu Q, Liu H, Meng S, Jiang T, Li X, Liang S, Ren S, Zhou C. First-line continual EGFR-TKI plus local ablative therapy demonstrated survival benefit in EGFR-mutant NSCLC patients with oligoprogressive disease. J Cancer. 2019 Jan 1;10(2):522-529. doi: 10.7150/jca.26494. eCollection 2019. PMID 30719148
- [Background] Qiu B, Liang Y, Li Q, Liu G, Wang F, Chen Z, Liu M, Zhao M, Liu H. Local Therapy for Oligoprogressive Disease in Patients With Advanced Stage Non-small-cell Lung Cancer Harboring Epidermal Growth Factor Receptor Mutation. Clin Lung Cancer. 2017 Nov;18(6):e369-e373. doi: 10.1016/j.cllc.2017.04.002. Epub 2017 Apr 12. PMID 28465010
- [Background] Iyengar P, Kavanagh BD, Wardak Z, Smith I, Ahn C, Gerber DE, Dowell J, Hughes R, Abdulrahman R, Camidge DR, Gaspar LE, Doebele RC, Bunn PA, Choy H, Timmerman R. Phase II trial of stereotactic body radiation therapy combined with erlotinib for patients with limited but progressive metastatic non-small-cell lung cancer. J Clin Oncol. 2014 Dec 1;32(34):3824-30. doi: 10.1200/JCO.2014.56.7412. Epub 2014 Oct 27. PMID 25349291
- [Background] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Petrakova K, Blackwell KL, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Mondal S, Su F, Miller M, Elmeliegy M, Germa C, O'Shaughnessy J. Updated results from MONALEESA-2, a phase III trial of first-line ribociclib plus letrozole versus placebo plus letrozole in hormone receptor-positive, HER2-negative advanced breast cancer. Ann Oncol. 2018 Jul 1;29(7):1541-1547. doi: 10.1093/annonc/mdy155. PMID 29718092
- [Background] Tripathy D, Im SA, Colleoni M, Franke F, Bardia A, Harbeck N, Hurvitz SA, Chow L, Sohn J, Lee KS, Campos-Gomez S, Villanueva Vazquez R, Jung KH, Babu KG, Wheatley-Price P, De Laurentiis M, Im YH, Kuemmel S, El-Saghir N, Liu MC, Carlson G, Hughes G, Diaz-Padilla I, Germa C, Hirawat S, Lu YS. Ribociclib plus endocrine therapy for premenopausal women with hormone-receptor-positive, advanced breast cancer (MONALEESA-7): a randomised phase 3 trial. Lancet Oncol. 2018 Jul;19(7):904-915. doi: 10.1016/S1470-2045(18)30292-4. Epub 2018 May 24. PMID 29804902
- [Background] Goetz MP, Toi M, Campone M, Sohn J, Paluch-Shimon S, Huober J, Park IH, Tredan O, Chen SC, Manso L, Freedman OC, Garnica Jaliffe G, Forrester T, Frenzel M, Barriga S, Smith IC, Bourayou N, Di Leo A. MONARCH 3: Abemaciclib As Initial Therapy for Advanced Breast Cancer. J Clin Oncol. 2017 Nov 10;35(32):3638-3646. doi: 10.1200/JCO.2017.75.6155. Epub 2017 Oct 2. PMID 28968163
- [Background] Johnston S, Martin M, Di Leo A, Im SA, Awada A, Forrester T, Frenzel M, Hardebeck MC, Cox J, Barriga S, Toi M, Iwata H, Goetz MP. MONARCH 3 final PFS: a randomized study of abemaciclib as initial therapy for advanced breast cancer. NPJ Breast Cancer. 2019 Jan 17;5:5. doi: 10.1038/s41523-018-0097-z. eCollection 2019. PMID 30675515
- [Background] Turner NC, Slamon DJ, Ro J, Bondarenko I, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Andre F, Puyana Theall K, Huang X, Giorgetti C, Huang Bartlett C, Cristofanilli M. Overall Survival with Palbociclib and Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2018 Nov 15;379(20):1926-1936. doi: 10.1056/NEJMoa1810527. Epub 2018 Oct 20. PMID 30345905
- [Background] Sledge GW Jr, Toi M, Neven P, Sohn J, Inoue K, Pivot X, Burdaeva O, Okera M, Masuda N, Kaufman PA, Koh H, Grischke EM, Frenzel M, Lin Y, Barriga S, Smith IC, Bourayou N, Llombart-Cussac A. MONARCH 2: Abemaciclib in Combination With Fulvestrant in Women With HR+/HER2- Advanced Breast Cancer Who Had Progressed While Receiving Endocrine Therapy. J Clin Oncol. 2017 Sep 1;35(25):2875-2884. doi: 10.1200/JCO.2017.73.7585. Epub 2017 Jun 3. PMID 28580882
- [Background] Slamon DJ, Neven P, Chia S, Fasching PA, De Laurentiis M, Im SA, Petrakova K, Bianchi GV, Esteva FJ, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Pivot X, Sondhi M, Wang Y, Chakravartty A, Rodriguez-Lorenc K, Taran T, Jerusalem G. Overall Survival with Ribociclib plus Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2020 Feb 6;382(6):514-524. doi: 10.1056/NEJMoa1911149. Epub 2019 Dec 11. PMID 31826360
- [Background] Xu B, Zhang Q, Zhang P, Hu X, Li W, Tong Z, Sun T, Teng Y, Wu X, Ouyang Q, Yan X, Cheng J, Liu Q, Feng J, Wang X, Yin Y, Shi Y, Pan Y, Wang Y, Xie W, Yan M, Liu Y, Yan P, Wu F, Zhu X, Zou J; DAWNA-1 Study Consortium. Dalpiciclib or placebo plus fulvestrant in hormone receptor-positive and HER2-negative advanced breast cancer: a randomized, phase 3 trial. Nat Med. 2021 Nov;27(11):1904-1909. doi: 10.1038/s41591-021-01562-9. Epub 2021 Nov 4. PMID 34737452
- [Background] Perey L, Paridaens R, Hawle H, Zaman K, Nole F, Wildiers H, Fiche M, Dietrich D, Clement P, Koberle D, Goldhirsch A, Thurlimann B. Clinical benefit of fulvestrant in postmenopausal women with advanced breast cancer and primary or acquired resistance to aromatase inhibitors: final results of phase II Swiss Group for Clinical Cancer Research Trial (SAKK 21/00). Ann Oncol. 2007 Jan;18(1):64-69. doi: 10.1093/annonc/mdl341. Epub 2006 Oct 9. PMID 17030543
- [Background] Johnston SR, Kilburn LS, Ellis P, Dodwell D, Cameron D, Hayward L, Im YH, Braybrooke JP, Brunt AM, Cheung KL, Jyothirmayi R, Robinson A, Wardley AM, Wheatley D, Howell A, Coombes G, Sergenson N, Sin HJ, Folkerd E, Dowsett M, Bliss JM; SoFEA investigators. Fulvestrant plus anastrozole or placebo versus exemestane alone after progression on non-steroidal aromatase inhibitors in postmenopausal patients with hormone-receptor-positive locally advanced or metastatic breast cancer (SoFEA): a composite, multicentre, phase 3 randomised trial. Lancet Oncol. 2013 Sep;14(10):989-98. doi: 10.1016/S1470-2045(13)70322-X. Epub 2013 Jul 29. PMID 23902874
- [Background] Martin JM, Handorf EA, Montero AJ, Goldstein LJ. Systemic Therapies Following Progression on First-line CDK4/6-inhibitor Treatment: Analysis of Real-world Data. Oncologist. 2022 Jun 8;27(6):441-446. doi: 10.1093/oncolo/oyac075. PMID 35552450
- [Background] Redig AJ, McAllister SS. Breast cancer as a systemic disease: a view of metastasis. J Intern Med. 2013 Aug;274(2):113-26. doi: 10.1111/joim.12084. PMID 23844915
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Griffioen G, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Bauman GS, Warner A, Senan S. Stereotactic ablative radiotherapy versus standard of care palliative treatment in patients with oligometastatic cancers (SABR-COMET): a randomised, phase 2, open-label trial. Lancet. 2019 May 18;393(10185):2051-2058. doi: 10.1016/S0140-6736(18)32487-5. Epub 2019 Apr 11. PMID 30982687
- [Background] Leone BA, Leone J, Leone JP. Breast cancer is a systemic disease rather than an anatomical process. Breast Cancer Res Treat. 2017 Feb;161(3):619. doi: 10.1007/s10549-017-4104-0. Epub 2017 Jan 9. No abstract available. PMID 28070768
- [Background] Leone BA, Vallejo CT, Romero AO, Machiavelli MR, Perez JE, Leone J, Leone JP. Prognostic impact of metastatic pattern in stage IV breast cancer at initial diagnosis. Breast Cancer Res Treat. 2017 Feb;161(3):537-548. doi: 10.1007/s10549-016-4066-7. Epub 2016 Dec 14. PMID 27975154
- [Background] Fisher B. The evolution of paradigms for the management of breast cancer: a personal perspective. Cancer Res. 1992 May 1;52(9):2371-83. No abstract available. PMID 1568206
- [Background] Loi M, Alifano M, Scorsetti M, Nuyttens JJ, Livi L. Judging a Fish by Its Ability to Climb a Tree? A Call for Novel Endpoints in the Appraisal of Ablative Local Treatments of Oligometastatic Cancer. Oncologist. 2021 Jun;26(6):e1085-e1086. doi: 10.1002/onco.13747. Epub 2021 Apr 9. PMID 33686724
- [Background] Buglione M, Jereczek-Fossa BA, Bonu ML, Franceschini D, Fodor A, Zanetti IB, Gerardi MA, Borghetti P, Tomasini D, Di Muzio NG, Oneta O, Scorsetti M, Franzese C, Romanelli P, Catalano G, Dell'Oca I, Beltramo G, Ivaldi GB, Laudati A, Magrini SM, Antognoni P; Italian Society of Radiotherapy and Clinical Oncology - Regional Group Lombardy (AIROL). Radiosurgery and fractionated stereotactic radiotherapy in oligometastatic/oligoprogressive non-small cell lung cancer patients: Results of a multi-institutional series of 198 patients treated with "curative" intent. Lung Cancer. 2020 Mar;141:1-8. doi: 10.1016/j.lungcan.2019.12.019. Epub 2020 Jan 3. PMID 31926440
- [Background] Klemen ND, Wang M, Feingold PL, Cooper K, Pavri SN, Han D, Detterbeck FC, Boffa DJ, Khan SA, Olino K, Clune J, Ariyan S, Salem RR, Weiss SA, Kluger HM, Sznol M, Cha C. Patterns of failure after immunotherapy with checkpoint inhibitors predict durable progression-free survival after local therapy for metastatic melanoma. J Immunother Cancer. 2019 Jul 24;7(1):196. doi: 10.1186/s40425-019-0672-3. PMID 31340861
- [Background] Sindhu KK, Leiter A, Moshier E, Lin JY, Carroll E, Brooks D, Shimol JB, Eisenberg E, Gallagher EJ, Stock RG, Galsky MD, Buckstein M. Durable disease control with local treatment for oligoprogression of metastatic solid tumors treated with immune checkpoint blockade. Cancer Treat Res Commun. 2020;25:100216. doi: 10.1016/j.ctarc.2020.100216. Epub 2020 Oct 8. PMID 33049542
- [Background] Desideri I, Francolini G, Scotti V, Pezzulla D, Becherini C, Terziani F, Delli Paoli C, Olmetto E, Visani L, Meattini I, Greto D, Bonomo P, Loi M, Detti B, Livi L. Benefit of ablative versus palliative-only radiotherapy in combination with nivolumab in patients affected by metastatic kidney and lung cancer. Clin Transl Oncol. 2019 Jul;21(7):933-938. doi: 10.1007/s12094-018-02005-7. Epub 2018 Dec 18. PMID 30565084
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774